CLINICAL TRIAL: NCT06347016
Title: Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Plozsiran in Adults With Severe Hypertriglyceridemia
Brief Title: Study of Plozasiran in Adults With Severe Hypertriglyceridemia
Acronym: SHASTA-4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROAPOC3-3004; 2023-509301-80 (EudraCT Number)
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — plozasiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Plozasiran Injection (Experimental): 4 doses of plozasiran (ARO-APOC3) by subcutaneous (sc) injection
  Interventions: Drug: Plozasiran Injection
- Placebo (Placebo Comparator): calculated volume to match active treatment by sc injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Plozasiran Injection — ARO-APOC3 Injection
  Other Names: ARO-APOC3
  Arms: Plozasiran Injection
Drug: Placebo — sterile normal saline (0.9% NaCl)
  Arms: Placebo

SUMMARY:
This Phase 3 study will evaluate the safety and efficacy of plozasiran injection (ARO-APOC3) in adult participants with severe hypertriglyceridemia (SHTG). After providing informed consent eligible participants will be randomized to receive 4 doses (once every 3 months) of plozasiran or placebo, and be evaluated for efficacy and safety. After Month 12, eligible participants will be offered an opportunity to continue in an optional open-label extension under a separate protocol.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of severe hypertriglyceridemia (SHTG) and prior documented evidence (medical history) of fasting TG levels of ≥500 mg/dL (≥5.65 mmol/L)
* Mean fasting TG level ≥500 mg/dL (≥5.65 mmol/L) collected at 2 separate and consecutive visits at least 7 days apart and no more than 17 days apart during the screening period
* Fasting low density lipoprotein-cholesterol (LDL-C) ≤130 mg/dL (≤3.37 mmol/L) at screening
* Screening HbA1C ≤9.0%
* Must be on standard of care lipid-lowering medications per local guidelines (unless documented as intolerant as determined by the Investigator, including an inability to safely administer or re-administer a specific drug because of fear, preference, genetic, clinical, or metabolic considerations, or due to a previous adverse reaction associated with, attributed to, or caused by specific drug)

Exclusion Criteria:

* Use of any hepatocyte-targeted small interfering ribonucleic acid (siRNA) that targets lipids and/or triglycerides within 365 days before Day 1 (except inclisiran, which is permitted). Administration of investigational drug and inclisiran must be separated by at least 4 weeks
* Use of any other hepatocyte-targeted siRNA or antisense oligonucleotide molecule within 60 days or within 5-half-lives before Day 1 based on plasma pharmacokinetics (PK), whichever is longer (except inclisiran, which is permitted)
* Known diagnosis of familial chylomicronemia syndrome (FCS) (type 1 Hyperlipoproteinemia) by documentation of confirmed homozygote or double heterozygote for loss-of-function mutations in type 1- causing genes
* Body mass index >45kg/m^2

Note: Additional Inclusion/Exclusion criteria may apply per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent change in fasting serum TG levels from baseline to Month 12 compared to placebo | Baseline, Month 12

SECONDARY OUTCOMES:
Percent Change in Fasting Serum TG Levels from Baseline to Month 10 Compared to Placebo | Baseline, Month 10
Proportion of subjects who achieve fasting TG levels of <500 mg/dL (<5.65 mmol/L) at Month 12 compared to placebo | Baseline, Month 12
Proportion of Subjects Who Achieve Fasting TG Levels of < 150 mg/dL (<1.69 mmol/L) at Month 12 compared to placebo | Baseline, Month 12
Percent change in remnant cholesterol (VLDL-C) from baseline to Month 12 compared to placebo | Baseline, Month 12
Percent change in non-HDL-C from baseline to Month 12 compared to placebo | Baseline, Month 12
Adjudicated AP Event Rate During the Treatment Period Compared to Placebo From Day 1 to Month 12 | Month 12
Number of Subjects with Adverse Events (AEs) and Serious Adverse Events (SAEs) Over Time through Month 12 as Compared to Placebo | From first dose of study drug through Month 12
Incidence Rates of New-Onset Diabetes Mellitus (NODM) Throughout the Course of Treatment | From first dose of study drug through Month 12
Incidence Rates of Impaired Glucose Tolerance Throughout the Course of Treatment | From first dose of study drug through Month 12
Incidence Rates of Worsening of Existing Diabetes Throughout the Course of Treatment | From first dose of study drug through Month 12
Change from Baseline in Hemoglobin A1c (HbA1c) and Other Glycemic Control Parameters During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Change from Baseline in Fasting Blood Glucose During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Change from Baseline in C-Peptide During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Change from Baseline in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Change from Baseline in Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related Adverse Events (TRAEs) Associated with Worsening Glycemic Control During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Initiation of New Medication for Hyperglycemia among Study Participants Not Known to Have Pre-existing Diabetes Mellitus During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Adjudicated Major Adverse Cardiovascular Events (MACE) Rates During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Incidence of Anti-drug Antibodies (ADA) to Plozasiran in Subjects Receiving Plozasiran Over Time Through Month 12 | From first dose of study drug through Month 12
Titers of Anti-drug Antibodies (ADA) to Plozasiran in Subjects Receiving Plozasiran Over Time Through Month 12 | From first dose of study drug through Month 12

CONTACTS AND LOCATIONS:
Locations (149):
- United States (50):
  - Research Site 1, Birmingham, Alabama
  - Research Site 2, Mobile, Alabama
  - Research Site 3, Beverly Hills, California
  - Research Site 4, Canoga Park, California
  - Research Site 5, Huntington Beach, California
  - Research Site 6, Lincoln, California
  - Research Site 7, Long Beach, California
  - Research Site 8, Oxnard, California
  - Research Site 9, Clearwater, Florida
  - Research Site 10, North Miami, Florida
  - Research Site 11, Sarasota, Florida
  - Research Site 12, Lawrenceville, Georgia
  - Research Site 13, Sugar Hill, Georgia
  - Research Site 14, Elkhart, Indiana
  - Research Site 15, Indianapolis, Indiana
  - Research Site 16, South Bend, Indiana
  - Research Site 17, Overland Park, Kansas
  - Research Site 18, Topeka, Kansas
  - Research Site 19, Metairie, Louisiana
  - Research Site 20, Annapolis, Maryland
  - Research Site 21, Jackson, Mississippi
  - Research Site 22, Fremont, Nebraska
  - Research Site 23, Norfolk, Nebraska
  - Research Site 24, Morristown, New Jersey
  - Research Site 26, New York, New York
  - Research Site 27, Riverhead, New York
  - Research Site 25, The Bronx, New York
  - Research Site 28, Asheboro, North Carolina
  - Research Site 29, Wilmington, North Carolina
  - Research Site 30, Beavercreek, Ohio
  - Research Site 31, Columbus, Ohio
  - Research Site 32, Oklahoma City, Oklahoma
  - Research Site 33, Horsham, Pennsylvania
  - Research Site 34, Newport, Pennsylvania
  - Research Site 35, Philadelphia, Pennsylvania
  - Research Site 36, Philadelphia, Pennsylvania
  - Research Site 37, Fort Mill, South Carolina
  - Research Site 38, Greenville, South Carolina
  - Research Site 39, Chattanooga, Tennessee
  - Research Site 40, Fort Worth, Texas
  - Research Site 41, Houston, Texas
  - Research Site 42, Houston, Texas
  - Research Site 43, Houston, Texas
  - Research Site 44, Sugar Land, Texas
  - Research Site 45, Tomball, Texas
  - Research Site 46, Victoria, Texas
  - Research Site 47, Bountiful, Utah
  - Research Site 48, St. George, Utah
  - Research Site 49, Manassas, Virginia
  - Research Site 50, Roanoke, Virginia
- Argentina (5):
  - Research Site 52, CABA, Buenos Aires
  - Research Site 51, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Research Site 54, Córdoba, Córdoba Province
  - Research Site 53, Godoy Cruz, Mendoza Province
  - Research Site 55, Rosario, Santa Fe Province
- Brazil (8):
  - Research Site 61, Salvador, Estado de Bahia
  - Research Site 56, Brasília, Federal District
  - Research Site 59, Belo Horizonte, Minas Gerais
  - Research Site 62, Aracaju, Sergipe
  - Research Site 57, Campinas, São Paulo
  - Research Site 58, Santo André, São Paulo
  - Research Site 60, São José do Rio Preto, São Paulo
  - Research Site 63, Recife
- Bulgaria (14):
  - Research Site 64, Byala
  - Research Site 65, Dimitrovgrad
  - Research Site 66, Haskovo
  - Research Site 67, Kyustendil
  - Research Site 68, Rousse
  - Research Site 69, Sevlievo
  - Research Site 76, Sofia
  - Research Site 70, Sofia
  - Research Site 73, Sofia
  - Research Site 71, Sofia
  - Research Site 75, Sofia
  - Research Site 72, Sofia
  - Research Site 74, Sofia
  - Research Site 77, Stara Zagora
- Canada (5):
  - Research Site 78, North Vancouver, British Columbia
  - Research Site 79, Chicoutimi, Quebec
  - Research Site 80, Laval, Quebec
  - Research Site 81, Québec, Quebec
  - Research Site 82, Terrebonne, Quebec
- Czechia (7):
  - Research Site 83, Brno
  - Research Site 84, Náchod
  - Research Site 85, Olomouc
  - Research Site 86, Prague
  - Research Site 88, Slaný
  - Research Site 89, Teplice
  - Research Site 87, Trutnov
- France (5):
  - Research Site 91, Marseille, Bouches-du-Rhône
  - Research Site 92, Pessac, Gironde
  - Research Site 93, Bayonne, Pyrenees Atlantiques
  - Research Site 94, Lyon, Rhone
  - Research Site 90, Paris
- Germany (4):
  - Research Site 95, Deggingen, Baden-Wurttemberg
  - Research Site 96, Wallerfing, Bavaria
  - Research Site 97, Magdeburg, Saxony-Anhalt
  - Research Site 98, Berlin, State of Berlin
- Hungary (6):
  - Research Site 99, Békéscsaba
  - Research Site 100, Kaposvár
  - Research Site 101, Miskolc
  - Research Site 102, Pécs
  - Research Site 104, Pécs
  - Research Site 103, Zalaegerszeg
- Latvia (8):
  - Research Site 107, Daugavpils
  - Research Site 105, Daugavpils
  - Research Site 106, Daugavpils
  - Research Site 108, Kuldīga
  - Research Site 109, Riga
  - Research Site 110, Riga
  - Research Site 111, Riga
  - Research Site 112, Tukums
- Lithuania (6):
  - Research Site 115, Kaunas
  - Research Site 113, Kaunas
  - Research Site 114, Kaunas
  - Research Site 118, Šiauliai
  - Research Site 116, Vilnius
  - Research Site 117, Vilnius
- New Zealand (3):
  - Research Site 119, Christchurch
  - Research Site 120, New Plymouth
  - Research Site 121, Newtown
- Poland (9):
  - Research Site 122, Bydgoszcz
  - Research Site 123, Gdynia
  - Research Site 124, Katowice
  - Research Site 129, Lodz
  - Research Site 125, Malbork
  - Research Site 126, Szczecin
  - Research Site 130, Torun
  - Research Site 127, Wroclaw
  - Research Site 128, Zamość
- Slovakia (4):
  - Research Site 134, Bratislava
  - Research Site 131, Nové Zámky
  - Research Site 132, Prešov
  - Research Site 133, Rožňava
- South Africa (12):
  - Research Site 135, Centurion, Gauteng
  - Research Site 136, Krugersdorp, Gauteng
  - Research Site 137, Pretoria, Gauteng
  - Research Site 138, Durban, KwaZulu-Natal
  - Research Site 144, Cape Town, Western Cape
  - Research Site 139, Cape Town, Western Cape
  - Research Site 140, Cape Town, Western Cape
  - Research Site 143, Cape Town, Western Cape
  - Research Site 145, Cape Town, Western Cape
  - Research Site 146, Mossel Bay, Western Cape
  - Research Site 142, Plettenberg Bay, Western Cape
  - Research Site 141, Somerset West, Western Cape
- Spain (3):
  - Research Site 149, A Coruña, La Coruña
  - Research Site 147, Madrid
  - Research Site 148, Seville

IPD SHARING:
Plan to Share IPD: Undecided